CLINICAL TRIAL: NCT00166205
Title: A Single-Arm, Multi-Center Study of the Safety and Effectiveness of The Swedish Adjustable Gastric Band (SAGB) in the Treatment of Morbid Obesity
Brief Title: Safety and Effectiveness Study of The Swedish Adjustable Gastric Band (SAGB) in the Treatment of Morbid Obesity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sheryl Helsinger, Director, Clinical Operations
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CI-02-0006
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Results first posted 2008-12-11 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Obesity, Morbid
Keywords: Obesity, Morbid; Obesity; Body Weight
MeSH Terms: conditions — Obesity, Morbid; Obesity; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gastric Band (Experimental): Single-arm study, all subjects banded.
  Interventions: Device: Swedish Adjustable Gastric Band

INTERVENTIONS:
Device: Swedish Adjustable Gastric Band — Long term implantable device.
  Other Names: Realize Band

SUMMARY:
The purpose of this study is to determine whether the Swedish Adjustable Gastric Band (SAGB) is safe, and effective in achieving weight loss in patients with Morbid Obesity.

DETAILED DESCRIPTION:
Surgical treatment of morbidly obese patients is considered a reasonable option for achieving weight loss when more conservative measures, such as diet and exercise have failed. Not only can weight loss be achieved, but also reduction / resolution of a patient's co-morbidities associated with excess weight. Adjustable gastric banding provides a less invasive, reversible bariatric surgery option. The SAGB has been commercially available outside the United States for this indication since 1996. Commercial availability has led to extensive literature supporting the safety and effectiveness of the SAGB. Given the available literature, a prospective, single arm, multicenter, study in a heterogeneous population of morbidly obese subjects in the U.S. is being conducted.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend, follow and give signed informed consent;
* 18 to 60 years of age (inclusive);
* Five year history of morbid obesity;
* Body Mass Index (BMI) >40 kg/m2 and <55 kg/m2, or BMI >35 kg/m2 and <40 kg/m2 with one or more significant medical conditions related to obesity (co-morbid conditions of type 2 diabetes, hyperlipidemia, obstructive sleep apnea, hypertension, metabolic syndrome, or osteoarthritis of the hip or knee) for which the subject is being treated, and which are generally expected to be improved, reversed, or resolved by weight loss.
* 100 lbs. overweight or 1.5 times ideal weight;
* Documented failure of conservative, non-surgical means of weight reduction within one year prior to the Screening Visit, including failure of supervised diet, exercise and or behavior modification programs, and pharmacologic therapy;
* Willing to commit to significant lifestyle changes that include diet, eating, and exercise habits for the duration of the clinical trial;
* Able to commit to long-term follow-up, including band adjustment visits:
* Living within the contiguous U.S. and is within a 100 mile radius of the study center;
* Absence of significant psychopathology that could limit the subject's ability to understand the procedure, comply with medical, surgical, and/or behavioral recommendations, as documented during screening assessment;
* Agrees to refrain from any type of reconstructive surgery that would affect body weight such as abdominal lipoplasty or liposuction, mammoplasty, or removal of excess skin for the follow-up period following SAGB placement; and
* Candidate for surgical weight loss intervention (i.e., meets accepted health criteria for major surgery).

Exclusion Criteria:

* Women of childbearing potential who are not practicing an effective method of birth control or who are pregnant or lactating;
* Previous malabsorptive or restrictive procedures performed for the treatment of obesity;
* Documented history of drug and/or alcohol abuse within two years of the Screening Visit;
* History of impaired mental status including, but not limited to active substance abuse, a history of schizophrenia, borderline personality disorder, uncontrolled depression, suicidal attempts within the past two years or current suicidal tendencies or ideations;
* Presence of any of the following medical conditions;

  * Inflammatory diseases of the gastrointestinal tract, including severe intractable esophagitis, gastric ulceration, duodenal ulceration, or specific inflammation such as Crohn's disease that have been active within the past 10 years;
  * Congenital or acquired anomalies of the GI tract, including atresias or stenosis,
  * Severe cardiopulmonary disease or other serious organic disease that makes the subject a high-risk surgical candidate;
  * Uncontrolled hypertension;
  * Portal Hypertension;
  * Uncontrolled Diabetes Mellitus;
  * Chronic or acute upper gastrointestinal bleeding conditions, e.g. gastric or esophageal varices;
  * Cirrhosis;
  * Congenital or acquired intestinal telangiectasia;
  * Esophageal or gastric disorders including severe preoperative reflux, dysmotility, or Barrett's Esophagus;
  * Presence of hiatal hernia;
  * Prior surgery of the foregut including hiatal hernia repair or prior gastric surgery;
  * Chronic pancreatitis;
  * Immunocompromised such as that resulting from chronic oral steroid use, chemotherapeutic agents, or immune deficiency disorders;
  * Conditions that, in the opinion of the investigator, may jeopardize the subject's well-being and/or the soundness of this clinical study;
* History or presence of pre-existing autoimmune connective tissue disease, i.e., systemic lupus erythematosus or scleroderma;
* Presence of terminal illness with life expectancy <5 years;
* Use of prescription or over the counter weight reduction medications or supplements within one month of the Screening Visit and for the duration of study participation;
* Acute or chronic infection (localized or systemic);
* Known or suspected allergy to silicone or other materials contained in the Swedish Adjustable Gastric Band;
* History of intolerance to implanted devices;
* Not ambulatory; and
* Participation in another clinical trial within 8 weeks of the Screening Visit and for the duration of this trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 276 (Actual)
Dates: Start 2003-06; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Phillips, MD, Principal Investigator — Cedars Sinai
Locations (12):
- United States (12):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Scripps Clinic Medical Group, San Diego, California
  - US Bariatrics, Fort Lauderdale, Florida
  - Advanced Surgical Institute at Mercy Hospital, Miami, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Hamilton Medical Center - Weight Management, Dalton, Georgia
  - Weight Management Center, New Orleans, Louisiana
  - University of Minnesota, Minneapolis, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - CAREMAX Surgical, P.C., East Patchogue, New York
  - St. Luke's-Roosevelt Hospital Center, New York, New York
  - Surgical Consultants of San Antonio, San Antonio, Texas

REFERENCES:
- [Background] Phillips E; SAGB Study Group. Design and demography of the United States Swedish Adjustable Gastric Band trial: a 3-year prospective study. Surg Obes Relat Dis. 2008 May-Jun;4(3 Suppl):S63-72. doi: 10.1016/j.soard.2008.04.009. PMID 18501317
- [Result] Phillips E, Ponce J, Cunneen SA, Bhoyrul S, Gomez E, Ikramuddin S, Jacobs M, Kipnes M, Martin L, Marema RT, Pilcher J, Rosenthal R, Rubenstein R, Teixeira J, Trus T, Zundel N. Safety and effectiveness of Realize adjustable gastric band: 3-year prospective study in the United States. Surg Obes Relat Dis. 2009 Sep-Oct;5(5):588-97. doi: 10.1016/j.soard.2008.12.007. Epub 2009 Jan 18. PMID 19342314
- See also: PubMed Abstract 3-yr Results — http://www.ncbi.nlm.nih.gov/pubmed/?term=19342314
- See also: PubMed Abstract Design — http://www.ncbi.nlm.nih.gov/pubmed/?term=18501317

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at twelve U.S. sites representative of the intended use of the SAGB in terms of both the subject population and the medical community. Subjects were recruited from a wide, heterogeneous subject population. Dates of recruitment June, 2003 to November, 2003.
Pre-assignment Details: 405 Subjects were consented. 129 did not meet screening criteria. 276 subjects were enrolled and received the SAGB device.
Period: Overall Study
Arm/Group | Swedish Adjustable Gastric Band (SAGB)
Started | 276
Intervention - SAGB Surgery | 276
Completed | 228
Not Completed | 48

BASELINE CHARACTERISTICS:
Arm/Group | Swedish Adjustable Gastric Band (SAGB)
Number analyzed (Participants) | 276
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 276
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 216
  Male | 60
Region of Enrollment [Number; unit: participants]
  United States | 276
Mean Excess Body Weight [Mean (Standard Deviation); unit: Pounds] — Excess weight is computed as baseline weight minus Ideal weight. Ideal weight as provided in the 1983 Metropolitan Life Height and Weight Table using the upper limit of the midpoint range.
  Pounds | 130.0 (33.1)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects Who Had Adverse Events With the Swedish Adjustable Gastric Band (SAGB)
Description: Percent of device-related adverse events (AEs) and device malfunctions occurring in subjects implanted with the Swedish Adjustable Gastric Band from baseline throughout the three-year post-operative period.
Time Frame: 3 years
Population: Intent to Treat (ITT)
Measure: Number; unit: Percent of Subjects
Arm/Group | Swedish Adjustable Gastric Band (SAGB)
Number analyzed (Participants) | 276
Percent of Subjects | 69.6
Statistical Analysis 1: Comparison: Swedish Adjustable Gastric Band (SAGB); A sample size of 215, the adverse event (AE) rate at three years could be estimated with precision as determined by the interval half-width of approximately ± 7%; Test type: Superiority or Other; Percent of ITT subjects = 69.6, 95% CI [63.8 to 74.9]

2. Secondary Outcome: Changes in Excess Body Weight (EBW)
Description: Changes in excess body weight at 3-years post-operative minus baseline excess weight. Excess weight is computed as baseline weight minus Ideal weight. Ideal weight as provided in the 1983 Metropolitan Life Height and Weight Table using the upper limit of the midpoint range.
Time Frame: 3 years
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | Swedish Adjustable Gastric Band (SAGB)
Number analyzed (Participants) | 276
Pounds | 75.7 (39.8)
Statistical Analysis 1: Comparison: Swedish Adjustable Gastric Band (SAGB); Test type: Superiority or Other; Mean = 75.7, 95% CI [70.5 to 80.8], Standard Deviation 39.8

3. Secondary Outcome: Changes in Body Mass Index (BMI)
Description: Changes in Body Mass Index (BMI) at three-years post-operative minus baseline.
Time Frame: 3 years
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Swedish Adjustable Gastric Band (SAGB)
Number analyzed (Participants) | 276
kg/m2 | 35.7 (6.2)
Statistical Analysis 1: Comparison: Swedish Adjustable Gastric Band (SAGB); Test type: Superiority or Other; Mean = 35.7, 95% CI [34.9 to 36.5], Standard Deviation 6.2

4. Secondary Outcome: Change in Absolute Weight
Description: Absolute weight loss as measured on a standardized Tanita Scale (used at all sites) at three-years post-operative minus baseline.
Time Frame: 3 years
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | Swedish Adjustable Gastric Band (SAGB)
Number analyzed (Participants) | 276
Pounds | 51.3 (30.8)
Statistical Analysis 1: Comparison: Swedish Adjustable Gastric Band (SAGB); Test type: Superiority or Other; Mean = 51.3, 95% CI [47.6 to 54.9], Standard Deviation 45.8

5. Secondary Outcome: Changes in Quality of Life (QOL) Measures
Description: Changes in QOL measures at three-years post-operative minus baseline. SF-36 scores from 0-100 with higher scores representing better QOL.
Time Frame: 3 years
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Swedish Adjustable Gastric Band (SAGB)
Number analyzed (Participants) | 276
Units on a scale | 10.4 (10.3)
Statistical Analysis 1: Comparison: Swedish Adjustable Gastric Band (SAGB); Test type: Superiority or Other; Mean Difference (Net) = 10.4, 95% CI [9.2 to 11.7], Standard Deviation 10.3 — Value at 36 months minus value at baseline. Positive values indicate improved Quality of Life (QOL)

6. Secondary Outcome: Changes in Glycosylated Hemoglobin (HbA1c)
Description: Changes in glycosylated hemoglobin (HbA1c), from baseline to three-years post-operative.
Time Frame: 3 years
Measure: Mean (Standard Deviation); unit: Percent of total hemogloobin
Arm/Group | Swedish Adjustable Gastric Band (SAGB)
Number analyzed (Participants) | 276
Percent of total hemogloobin | 5.7 (0.7)
Statistical Analysis 1: Comparison: Swedish Adjustable Gastric Band (SAGB); Test type: Superiority or Other; Mean = 5.7, 95% CI [5.6 to 5.8], Standard Deviation 0.7

7. Secondary Outcome: Number of All Adverse Events of Subjects Implanted With the SAGB
Description: The evaluation of all Adverse Events of subjects implanted with the Swedish Adjustable Gastric Band throughout the three-year post-operative period (related to device and unrelated to device).
Time Frame: 3 Years
Measure: Number; unit: Total Number of Adverse Events
Arm/Group | Swedish Adjustable Gastric Band (SAGB)
Number analyzed (Participants) | 276
Total Number of Adverse Events | 2400

8. Primary Outcome: Percent Excess Weight Loss
Description: Percent Excess Weight Loss (%EWL) with the SAGB at three years post operatively minus baseline.
Time Frame: 3 Years Post Operative
Population: Intent to Treat (ITT), Last Observation Carried Forward (LOCF)
Measure: Mean (95% Confidence Interval); unit: Percent Excess Weight Loss
Arm/Group | Swedish Adjustable Gastric Band (SAGB)
Number analyzed (Participants) | 276
Percent Excess Weight Loss | 41.1 [38.1 to 44.1]
Statistical Analysis 1: Comparison: Swedish Adjustable Gastric Band (SAGB); A one-sided paired t-test would have 80% power to reject the null hypothesis in favor of the alternative (i.e., that the SAGB system is not inferior to the clinically meaningful result of 36.2 for 224 subjects) assuming: a standard deviation (SD) of (21.6), an equivalent limit difference of (3.6), and a significance level of 0.05; Test type: Superiority or Other; p < 0.001, t-test, 1 sided

9. Secondary Outcome: Changes in High Density Lipoproteins (HDL)
Description: Changes in High Density Lipoproteins (HDL), at three-years post-operative minus baseline.
Time Frame: 3 year
Measure: Mean (Standard Deviation); unit: Mg/dl
Arm/Group | Swedish Adjustable Gastric Band (SAGB)
Number analyzed (Participants) | 276
Mg/dl | 56.4 (14.7)
Statistical Analysis 1: Comparison: Swedish Adjustable Gastric Band (SAGB); Test type: Superiority or Other; Mean = 56.4, 95% CI [54.5 to 58.4], Standard Deviation 14.7

10. Secondary Outcome: Changes in Low Density Lipoproteins (LDL)
Description: Changes in Low Density Lipoproteins (LDL), at three-years post-operative minus baseline.
Time Frame: 3 years
Measure: Mean (Standard Deviation); unit: Mg/dl
Arm/Group | Swedish Adjustable Gastric Band (SAGB)
Number analyzed (Participants) | 276
Mg/dl | 114.5 (32.3)
Statistical Analysis 1: Comparison: Swedish Adjustable Gastric Band (SAGB); Test type: Superiority or Other; Mean = 114.5, 95% CI [110.1 to 118.8], Standard Deviation 32.3

11. Secondary Outcome: Changes in Total Cholesterol
Description: Changes in Total Cholesterol, at three-years post-operative minus baseline.
Time Frame: 3 years
Measure: Mean (Standard Deviation); unit: Mg/dl
Arm/Group | Swedish Adjustable Gastric Band (SAGB)
Number analyzed (Participants) | 276
Mg/dl | 193.5 (36.9)
Statistical Analysis 1: Comparison: Swedish Adjustable Gastric Band (SAGB); Test type: Superiority or Other; Mean = 193.5, 95% CI [188.6 to 198.4], Standard Deviation 36.9

ADVERSE EVENTS:
Time Frame: Date of surgery to 3 years post-surgery
Description: Subjects were questioned at all visits regarding any changes in their physical health.
Arm/Group | Swedish Adjustable Gastric Band (SAGB)
Serious Adverse Events (participants affected / at risk) | 78/276
Other Adverse Events (participants affected / at risk) | 266/276
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Swedish Adjustable Gastric Band (SAGB) (N=276)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiomegaly (Cardiac disorders) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Gastric dilatation (Gastrointestinal disorders) | 3 (3)
Gastric outlet obstruction (Gastrointestinal disorders) | 3 (3)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2)
Gastrointestinal oedema (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Oesophageal spasm (Gastrointestinal disorders) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Pancreatitis due to biliary obstruction (Gastrointestinal disorders) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3)
Catheter related complication (General disorders) | 14 (15)
Chest pain (General disorders) | 3 (3)
Drug withdrawal syndromwe (General disorders) | 1 (1)
Impaired healing (General disorders) | 1 (1)
Migration of implant (General disorders) | 15 (17)
Biliary colic (Hepatobiliary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 4 (4)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 5 (5)
Hypersensitivity (Immune system disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Injection site infection (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Device failure (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Gastrointestinal injury (Injury, poisoning and procedural complications) | 2 (2)
Injury (Injury, poisoning and procedural complications) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1)
Surgical procedure repeated (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute myeloid leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Benign intracranial hypertension (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 1 (1)
Lumbar spinal stenosis (Nervous system disorders) | 1 (1)
Syncope vasovagal (Nervous system disorders) | 1 (1)
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Vomiting in pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (2)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1)
Urethral disorder (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Fibrocystic breast disease (Reproductive system and breast disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary microemboli (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Swedish Adjustable Gastric Band (SAGB) (N=276)
Vomiting (Gastrointestinal disorders) | 123
Nausea (Gastrointestinal disorders) | 89
Constipation (Gastrointestinal disorders) | 67
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 52
Abdominal pain (Gastrointestinal disorders) | 28
Flatulence (Gastrointestinal disorders) | 28
Abdominal pain upper (Gastrointestinal disorders) | 27
Diarrhoea (Gastrointestinal disorders) | 26
Dysphagia (Gastrointestinal disorders) | 26
Dyspepsia (Gastrointestinal disorders) | 23
Fatigue (General disorders) | 29
Injection site pain (General disorders) | 18
Nasopharynigitis (Infections and infestations) | 30
Influenza (Infections and infestations) | 26
Sinusitis (Infections and infestations) | 22
Urinary tract infection (Infections and infestations) | 21
Upper respiratory tract infection (Infections and infestations) | 20
Post procedural pain (Injury, poisoning and procedural complications) | 66
Back pain (Musculoskeletal and connective tissue disorders) | 40
Arthralgia (Musculoskeletal and connective tissue disorders) | 27
Headache (Nervous system disorders) | 37
Depression (Psychiatric disorders) | 28
Insomnia (Psychiatric disorders) | 17
Alopecia (Skin and subcutaneous tissue disorders) | 24
Hypertension (Vascular disorders) | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI shall have the right to publish the results of research to include in any publication. The PI will provide the Sponsor with at least sixty (60) days for review of a manuscript. No paper that incorporates Sponsor Confidential Information will be submitted for publication without Sponsor's prior written agreement.